CLINICAL TRIAL: NCT02874768
Title: Comparison Between Dexmedetomidine and Propofol for Postoperative Sedation of Patients in the Intensive Care Unit After Abdominal Surgery: Microcirculation, Kidney Injury, and Intestinal Injury
Brief Title: Comparison Between Dexmedetomidine and Propofol for Patients in the Intensive Care Unit After Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201605038MINB
Record Dates: First submitted 2016-08-05; First posted 2016-08-22 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Microcirculation
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): Patient receives continuous intravenous infusion of dexmedetomidine (infusion dosage range: 0.1 ~ 0.7 mcg/kg/h)
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Patient receives continuous intravenous infusion of propofol (infusion dosage range: 0.3 ~ 1.6 mg/kg/h)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Patient receives continuous intravenous infusion of dexmedetomidine (infusion dosage range: 0.1 ~ 0.7 mcg/kg/h)
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: Propofol — Patient receives continuous intravenous infusion of propofol (infusion dosage range: 0.3 ~ 1.6 mg/kg/h)
  Other Names: Fresofol
  Arms: Propofol

SUMMARY:
This is a single-blind randomized clinical trial. Patients undergoing abdominal surgery will be enrolled and randomly divided into two groups: dexmedetomidine group and propofol group. In the dexmedetomidine group, patients will receive continuous intravenous infusion of dexmedetomidine (infusion dosage range: 0.1 ~ 0.7 mcg/kg/h). In the propofol group, patients will receive continuous intravenous infusion of propofol (infusion dosage range: 0.3 ~ 1.6 mg/kg/h). Hemodynamics will be continuously monitored using a non-invasive monitoring with chest bioreactance technique at preset time points (0, 2, 4, 6, 12h and 24h). Clinical data such as vital signs, hemodynamic parameters, laboratory results and fluid balance will be recorded. The microcirculation will be examined by Cytocam. The following microcirculatory parameters will be investigated: total small vessel density, perfused small vessel density, microvascular flow index, and heterogeneity index. The enzyme-linked immunosorbent assays will be used to measure serum level of endocan, diamine oxidase, and neutrophil gelatinase-associated lipocalin at preset time points. The primary goal of this study is to compare the effect on microcirculation between dexmedetomidine and propofol in intensive care unit patients after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* non-emergent major abdominal surgery with ICU admission
* the need of sedation during ICU stay

Exclusion Criteria:

* age younger than 20 years and older than 89 years
* refractory bradycardia (HR < 60 bpm after treatment)
* severe AV block (2nd or 3rd degree)
* refractory shock (MAP < 60 mm Hg after treatment)
* severe heart failure or NYHA 4
* new onset of myocardial infarction within 4 weeks
* receive CPR within 4 weeks
* APACHE score > 30 before enrollment
* severe liver cirrhosis or CHILD B or C
* pregnancy
* allergic history to dexmedetomidine or propofol
* be enrolled in other clinical trials related to dexmedetomidine or propofol within 4 weeks
* non-native speakers

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Total perfused small vessel density | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No